CLINICAL TRIAL: NCT04288336
Title: A Prospective Pilot Study Evaluating the Feasibility of Daily, Long-Term Intermittent Fasting for Men on PSA Surveillance Following Radical Prostatectomy for Localized, High-Risk Prostate Cancer
Brief Title: Daily, Long-Term Intermittent Fasting for the Prevention of PSA-Recurrence in Patients With Localized Prostate Cancer After Radical Prostatectomy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No patient accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-006675; NCI-2020-00832 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC2052; 19-006675 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (intermittent fasting) (Experimental): Beginning when patients' PSA is detectable up to 24 months after surgery, patients follow a daily intermittent fasting routine consisting of restricting the daily eating period to 8 hours (e.g. between 1PM-9PM) followed by 16 hours of prolonged nightly fasting for up to 1 year or until secondary therapy commences.
  Interventions: Other: Food Diary; Other: Preventative Dietary Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Food Diary — Ancillary studies
Other: Preventative Dietary Intervention — Follow intermittent fasting
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial studies the feasibility of a daily, long-term intermittent fasting routine in preventing or delaying a rise in prostate specific antigen (PSA) levels in patients with prostate cancer that has not spread to other parts of the body (localized) and who have undergone radical prostatectomy. PSA is a protein produced by both normal and cancer cells. Following a daily fasting routine after treatment for prostate cancer may lower the risk of patients' PSA level rising above 0.4 ng/mL, which is also called PSA-recurrence. A PSA-recurrence can sometimes mean that the disease has returned and/or progressed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether men treated for localized prostate cancer adhere to a long-term (months-years) daily intermittent fasting regimen.

II. To measure the levels of metabolic and prostate-cancer derived microparticles in the serum of men that practice a daily intermittent fasting regimen after treatment for localized, high-risk prostate cancer.

OUTLINE:

Beginning when patients' PSA is detectable up to 24 months after surgery, patients follow a daily intermittent fasting routine consisting of restricting the daily eating period to 8 hours (e.g. between 1PM-9PM) followed by 16 hours of prolonged nightly fasting for up to 1 year or until secondary therapy commences.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven histological diagnosis of localized prostate cancer (pT2 or specimen confined pT3)
* Having undergone radical prostatectomy (open or laparoscopic) with bilateral pelvic lymph node dissection
* Negative surgical margins on final specimen
* Men that decline adjuvant therapy
* Detectable serum PSA of 0.1 ng/mL or >
* 24 months or less since radical prostatectomy at time of study screening

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Treated prior to surgery with any form of hormone, antiandrogen, or androgen deprivation therapy
* Treated prior to surgery with any form of chemotherapy or radiotherapy
* Medical conditions/history that precludes subjects from following a fasting regimen, including but not limited to:

  * Diabetes mellitus
* On hormone therapy (Casodex, gonadotrophin releasing hormone [GnRH] agonist/antagonist)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Adherence to the daily intermittent fasting regimen | Up to 1 year
  Will be assessed via the phone surveys conducted at each remote follow up visit, as well as through analysis of the subjects' daily journals that will be sent back to the study team at the end of the study period.

SECONDARY OUTCOMES:
Prostate specific antigen (PSA) kinetics and/or doubling time | Up to 1 year
  Will assess the PSA kinetics and/or doubling time as it relates to historical patients whom have also undergone PSA surveillance with postoperative PSA detection 0.1 or >.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Karnes, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials